CLINICAL TRIAL: NCT00738218
Title: Coronary Evaluation Using Multi-Detector Spiral Computed Tomography Angiography Using 64 Detectors: "CORE-64" Study
Brief Title: Diagnostic Accuracy of Multi-Detector Spiral Computed Tomography Angiography Using 64 Detectors
Acronym: CORE-64
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Joao A. C. Lima, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: JHUCORE64; NA_00003755; NTR535
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Computed Tomography; Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDCT (Other): Single Arm study. All patients underwent MDCT.
  Interventions: Other: Multidetector Computed Tomography - 64 detectors

INTERVENTIONS:
Other: Multidetector Computed Tomography - 64 detectors — Multidetector computed tomography angiography
  Other Names: Aquillion 64 detector CT scanner

SUMMARY:
To compare the diagnostic ability of 64-detector MDCT coronary angiography with conventional invasive coronary angiography in patients with suspected coronary artery disease.

DETAILED DESCRIPTION:
The "Coronary Evaluation Using Multidetector Spiral Computed Tomography Angiography using 64 Detectors" or "CorE-64" study was designed to evaluate the diagnostic accuracy of multislice spiral CT angiography using 64 detector rows for identifying coronary artery stenosis in patients with suspected or known coronary artery disease. The study was designed as a prospective, multi-center, international, blinded study examining the diagnostic accuracy of 64-slice CT in comparison with CCA. The primary hypothesis of the study is that 64-slice CT coronary angiography will be able to detect significant coronary artery disease in a patient with acceptable diagnostic accuracy as compared to CCA. Significant CAD is defined as ≥ 50% stenosis as determined by quantitative analysis of CCA (QCA). The diagnostic parameters is per-patient sensitivity and specificity compared with CCA, with both point estimates and continuous measurements of diagnostic accuracy. Eligible patients will first undergo MDCT (calcium scanning and MDCTA)prior to clinically indicated conventional coronary angiography. Patients with CAC 600 or less will be included in the primary analysis. Patients will be followed for clinical events including revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 40 years or greater.
* Women of child bearing potential must demonstrate a negative pregnancy test within 24 hours of the study MDCT.
* Suspected coronary artery disease (i.e. symptoms, signs) with a clinical indication for coronary angiography; and planned coronary angiography within the next 30 days.
* Able to understand and willing to sign informed consent.

Exclusion Criteria:

* Known allergy to iodinated contrast media
* History of contrast-induced nephropathy
* History of multiple myeloma or previous organ transplantation
* Elevated serum creatinine (> 1.5mg/dl) OR calculated creatinine clearance of < 60 ml/min (using the Cockcroft-Gault formula
* Atrial fibrillation or uncontrolled tachyarrhythmia, or heart block
* Evidence of severe symptomatic heart failure; moderate or severe aortic stenosis
* Previous coronary artery bypass or other cardiac surgery
* Coronary artery intervention within the last 6 months
* Intolerance or contraindication to beta-blockers
* Body Mass Index > 40.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2005-10; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy to detect significant coronary artery disease in an individual patient. | 30 Days

SECONDARY OUTCOMES:
Diagnostic Accuracy to detect significant coronary artery disease in an individual vessel. | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Joao AC Lima, M.D., Principal Investigator — Johns Hopkins University; Julie M Miller, M.D., Principal Investigator — Johns Hopkins University; Joao AC Lima, M.D., Study Chair — Johns Hopkins University

REFERENCES:
- [Derived] Sara L, Rochitte CE, Lemos PA, Niinuma H, Dewey M, Shapiro EP, Gottlieb I, Mansur AP, Nicolau JC, Lardo AC, Azevedo CF, Kalil-Filho R, Vavere AL, Cohn S, Cox C, Brinker J, Miller JM, Lima JA. Accuracy of multidetector computed tomography for detection of coronary artery stenosis in acute coronary syndrome compared with stable coronary disease: a CORE64 multicenter trial substudy. Int J Cardiol. 2014 Dec 15;177(2):385-91. doi: 10.1016/j.ijcard.2014.08.130. Epub 2014 Aug 27. PMID 25281436
- [Derived] Yan RT, Miller JM, Rochitte CE, Dewey M, Niinuma H, Clouse ME, Vavere AL, Brinker J, Lima JA, Arbab-Zadeh A. Predictors of inaccurate coronary arterial stenosis assessment by CT angiography. JACC Cardiovasc Imaging. 2013 Sep;6(9):963-72. doi: 10.1016/j.jcmg.2013.02.011. Epub 2013 Aug 8. PMID 23932641
- [Derived] Gottlieb I, Miller JM, Arbab-Zadeh A, Dewey M, Clouse ME, Sara L, Niinuma H, Bush DE, Paul N, Vavere AL, Texter J, Brinker J, Lima JA, Rochitte CE. The absence of coronary calcification does not exclude obstructive coronary artery disease or the need for revascularization in patients referred for conventional coronary angiography. J Am Coll Cardiol. 2010 Feb 16;55(7):627-34. doi: 10.1016/j.jacc.2009.07.072. PMID 20170786
- [Derived] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879